CLINICAL TRIAL: NCT05292300
Title: Investigation of the Efficacy of Lyophilized Dried Cornelian Cherry (Cornus Mas L.) Fruit on Anthropometric and Biochemical Parameters in Women With Insulin Resistance
Brief Title: Efficacy of Lyophilized Dried Cornus Mas L. on Anthropometric and Biochemical Parameters in Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zehra Margot Celik, Nutrition and Dietetics, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2018.652
Record Dates: First submitted 2021-08-31; First posted 2022-03-23 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Insulin Resistance; Obesity; PreDiabetes
Keywords: Cornelian Cherry; Cornus mas L.; Insulin Resistance; Nutrition; Anthropometry
MeSH Terms: conditions — Insulin Resistance; Obesity; Prediabetic State | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Among those who applied to the clinic, those who do not want to follow their diet will be randomized into this group.
- Cornelian Cherry Group (Experimental): Among those who applied to the clinic, those who do not want to follow their diet will be randomized into this group. Patients in this group will receive 20 g/day Cornelian Cherry powder.
  Interventions: Dietary Supplement: Cornelian Cherry (Cornus mas L.)
- Diet Group (Experimental): Among those who applied to the clinic, those who want to follow their diet will be randomized into this group. Patients in this group will be followed by a personalized diet.
  Interventions: Behavioral: Diet
- Cornelian Cherry and Diet Group (Experimental): Among those who applied to the clinic, those who want to follow their diet will be randomized into this group. Patients in this group will be followed by a personalized diet and will receive 20 g/day Cornelian Cherry powder for their one portion fruit a day.
  Interventions: Dietary Supplement: Cornelian Cherry (Cornus mas L.); Behavioral: Diet

INTERVENTIONS:
Dietary Supplement: Cornelian Cherry (Cornus mas L.) — Patients in "Cornelian Cherry Group" and "Cornelian Cherry and Diet Group" will receive 20 g/day freeze-dried powder Cornelian Cherry supplement.
  Arms: Cornelian Cherry Group; Cornelian Cherry and Diet Group
Behavioral: Diet — Patient in "Diet Group" and "Cornelian Cherry and Diet Group" will be given a personalized diet and be followed up by a dietician.
  Arms: Cornelian Cherry and Diet Group; Diet Group

SUMMARY:
The aim of this study is to determine the effect of 3 months supplementation of lyophilize dried cornelian cherry (Cornus mas L.) on women diagnosed with insulin resistance. The baseline and end biochemical parameters and anthropometric measurements will be compared with control subjects.

DETAILED DESCRIPTION:
The main purpose of this study is to determine the efficacy of the lyophilizer-dried powder form of cornelian cherry (Cornus mas L.) grown in our country on inflammation in women with insulin resistance by biochemical parameters.

Sub-objectives of the study;

* Determining the presence of inflammation in women with insulin resistance.
* Determination of the effect of cornelian cherry on both fasting blood glucose, insulin and blood lipid profile.
* Determination of both anti-inflammatory, antidiabetic and antioxidant effects of cornelian cherry.
* Determination of the effect of cornelian cherry on anthropometric measurements.

The aim of this study is to compare the anthropometric measurements and biomarkers of women with insulin resistance as a result of the consumption of powdered cornelian cherry (Cornus mas L.) that has been freeze-dried at -55 degrees with a Lyophilizer device for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 45 years with insulin resistance.
* Those who have not experienced menopause
* Those who applied to the obesity clinic
* Volunteers
* Those who signed the consent form

Exclusion Criteria:

* Those who use medicine for diabetes and thyroid diseases,
* Those taking hormone therapy
* Pregnant and lactating women
* Those with a history of cancer
* Patients with communication problems.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Fasting Blood Glucose (mg/dl) at 12 weeks | 3 months
  The fasting blood glucose (mg/dl) at the baseline and 12 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 3 months), Cornelian Cherry and Diet Group (who received additional 20 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 20 g/day of dried powdered Cornelian Cherry ).
Change from Baseline in the Fasting Insulin (mU/L) at 12 weeks | 3 months
  The fasting insulin (mU/L) values of the women with insulin resistance at the baseline and 12 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 3 months), Cornelian Cherry and Diet Group (who received additional 20 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 20 g/day of dried powdered Cornelian Cherry ).
Change from Baseline in the HOMA-IR at 12 weeks | 3 months
  The fasting blood glucose (mg/dl) and fasting insulin (mU/L) values of the women with insulin resistance at the baseline and 12 weeks later will be taken noted from the routinely requested tests in the hospital. HOMA-IR will be calculated with the formula (fasting glucose (mg/dl) x fasting insulin (mU/L)) / 405. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 3 months), Cornelian Cherry and Diet Group (who received additional 20 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 20 g/day of dried powdered Cornelian Cherry ).
Change from Baseline in the BMI (kg/m2) | 3 months
  The body weight (kg) and height (m) of the women with insulin resistance at the baseline, 4 weeks, 8 weeks and 12 weeks will be taken by the researcher and noted in their files.
  The height of the patients will be measured with a fixed height meter with 0.5 cm intervals, with shoes off.
  For body analysis, an 8-electrode bioelectrical impedance (BIA) device Tanita MC 780 MA, which performs segmental analysis, will be used. Patients will be asked to remove all metal items (rings, earrings, bracelets, watches, phones, etc.), any heavy clothing, shoes, and socks before stepping on the device. The device is set to -1.0 kg for the remaining clothes.
  From these measurements, body weight, body fat (kg), body fat percentage (%), body muscle (kg) and body water (kg) values will be recorded. Body mass index (BMI) will be calculated as weight (kg) divided by height (m) squared.
Change from Baseline in the Anthropometric Measurements | 3 months
  The anthropometric measurements of the women with insulin resistance at the baseline, 4, 8 and 12 weeks will be taken by the researcher. These measurements are; waist circumference(cm), hip circumference(cm), mid-upper arm circumference(cm), neck circumference(cm), waist to height ratio(cm) and waist to hip ratio(cm). Waist circumference will be measured using an inflexible tape at the umbilicus level after normal exhalation to the nearest 0-1 cm. Hip circumference will be measured from the widest area between the waist and the thigh. The waist-to-hip will be calculated from the formula waist(cm)/hip(cm) and waist-to-height ratios will be calculated from the formula waist(cm)/height(cm). Middle-upper arm circumference will be measured on the left arm of the patients. Neck circumference will be measured with the shoulders in the free position from the point where the thyroid cartilage is most protruding.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Esra Güneş, PhD, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No